CLINICAL TRIAL: NCT05895227
Title: Hemorrhagic Complications of Transvaginal Oocyte's Retrieval: an Update.
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 16/23
Record Dates: First submitted 2023-03-14; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: ART; Infertility
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Oocyte retrieval

SUMMARY:
The goal of this retrospective analysis is to focus on peritoneal bleeding after oocyte retrieval and to further investigate factors related to this specific complication and if hemorrhagic complication rate modifications can be observed.

DETAILED DESCRIPTION:
The main aim is to update our knowledge on oocyte retrieval complication, focusing specifically on hemorrhagic / hemoperitoneum rate.

All retrievals will be retrieved in IVF/ICSI cycles and Fertility Preservation both in oncological patients and in patients requesting oocyte storage for deferring motherhood.

Data collection goes from January 2017 to December 2022.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent a procedure of oocyte transvaginal retrieval for IVF/ intracytoplasmatic sperm injection (ICSI) cycles and fertility preservation

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients that underwent oocyte retrieval procedure at Humanitas Fertility Center during the period January 2017 - December 2022, in IVF/ICSI cycles and fertility preservation both in oncological patients and in patients requesting oocyte storage for deferring motherhood.
Sampling Method: Probability Sample
Enrollment: 13193 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Hemoperitoneum after oocyte transvaginal retrieval | Oocyte retrievals in the period January 2017- December 2022
  number of patients with onset of hemoperitoneum

SECONDARY OUTCOMES:
Operator of the procedure | 6 years
  assessment of operator experience
Hemoglobin level before and after procedure | 6 years
  evaluation of hemoglobin level before and the day after procedure
Time of symptoms onset | 6 years
  evaluation of first symptoms onset
Loss of blood during procedure | 6 years
  average blood loss
Incidence compared to past case history | 6 years
  comparison with previous statistic
Need for hospitalization | 6 years
  patients requiring hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Emanuele Levi Setti, M.D., Principal Investigator — Istituto Clinico Humanitas